CLINICAL TRIAL: NCT01765660
Title: Mesenchymal Stem Cells From Third-party Donors for Treatment of Refractory Chronic Graft-versus-host Disease
Brief Title: Mesenchymal Stem Cells for Treatment of Refractory Chronic Graft-versus-host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-sen University (Other); Peking University People's Hospital (Other); Guangdong Provincial People's Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Southern Medical University, China (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFH-MSCs-cGVHD-2013
Record Dates: First submitted 2013-01-05; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: Hematopoietic Stem Cell Transplantation; Mesenchymal Stem Cells; Chronic Graft-versus-host disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-mesenchymal stem cells (Experimental): Non-mesenchymal stem cell group refers to treatment with other second line drugs
  Interventions: Biological: Non-mesenchymal stem cells
- Mesenchymal stem cells (Experimental): Mesenchymal stem cell group refers to treatment with mesenchymal stem cells (1×10^6 cells/kg, intravenously)every two weeks, four times for a cycle
  Interventions: Biological: Mesenchymal stem cells

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal stem cells will be intravenously infused via a central venous catheter(at a dose of 1×10^6 cells/kg, over 15 mins) every two weeks, four times for a cycle.
  Other Names: MSCs
  Arms: Mesenchymal stem cells
Biological: Non-mesenchymal stem cells — Other second line drugs are taken.
  Other Names: Non-MSCs
  Arms: Non-mesenchymal stem cells

SUMMARY:
The purpose of this study is to evaluate the utility of treating patients experiencing refractory chronic graft-versus-host disease with ex-vivo-expanded BM-drived mesenchymal stem cells from third-party donors. The objective was to evaluate the effect and safety of such treatment on refractory chronic graft-versus-host disease.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation(allo-HSCT) can cure many hematologic diseases. Although great progress has been made in the prevention and treatment of side effects associated with transplantation,chronic graft-versus-host disease(cGVHD) remains an important complication that occurs in about 50% patients. The mortality of cGVHD and its complication could reach up to 50%,and cGVHD seriously influence the quality of life. At present, glucocorticoids and cyclosporine (CsA) are the first line treatment of cGVHD, but their effective rates are only 50%. If first line treatment is ineffective, second line drugs would be taken, such as mycophenolate mofetil(MMF)and rituximab. The effective rates of second line drugs are 30%-61%. The effective rates and prognosis of refractory cGVHD are even worse.

Mesenchymal stem cells (MSCs) are a form of multipotent adult stem cells that can be isolated from bone marrow (BM), adipose tissue, and cord blood. Clinical applications of human MSCs are evolving rapidly with goals of improving hematopoietic engraftment, preventing and treating GVHD after allo-HSCT and so on. However, the efficacy of treatment of refractory cGVHD using expanded BM-derived MSCs from a third-party donor is rarely reported. If such treatment could be shown to be effective and safe, BM-derived MSCs could potentially be used as an universal donor material. This would have a major impact because the generation of donor-specific MSCs is time-consuming, costly, and often impractical if the clinical status of a patient is urgent.

In the present study, the investigators will prospectively evaluate the efficacy and safety of ex-vivo-expanded BM-derived MSCs from third-party donors in treating patients with refractory cGVHD.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 12-65 years
* Recipients of allogeneic hematopoietic stem cell transplantation
* Patients with refractory cGVHD
* On a voluntary basis, patients are divided into MSCs and Non-MSCs group
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of treatment for refractory cGVHD | 1 year
  The response criteria include complete response (CR), part response (PR), stable disease(SD) and progressive disease(PD). CR:cGVHD symptoms and signs disappear; PR:cGVHD symptoms and signs improve; SD:cGVHD symptoms and signs remain (without improvement or deterioration);PD: cGVHD symptoms and signs deteriorate.

SECONDARY OUTCOMES:
acute and late toxic side effects of MSCs treatment | 1 year
  Toxic side effects of treatment includes acute toxicity and late side effects. Acute toxicity principally involves the heart,live and kidney. Late toxic side effects involves principally the development of secondary tumors and relapse of the primary disease.

OTHER OUTCOMES:
infections | 1 year
  Infections will be mainly focused within the first 100 days after MSCs treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Perez-Simon JA, Lopez-Villar O, Andreu EJ, Rifon J, Muntion S, Diez Campelo M, Sanchez-Guijo FM, Martinez C, Valcarcel D, Canizo CD. Mesenchymal stem cells expanded in vitro with human serum for the treatment of acute and chronic graft-versus-host disease: results of a phase I/II clinical trial. Haematologica. 2011 Jul;96(7):1072-6. doi: 10.3324/haematol.2010.038356. Epub 2011 Mar 10. PMID 21393326
- [Background] Ringden O, Uzunel M, Rasmusson I, Remberger M, Sundberg B, Lonnies H, Marschall HU, Dlugosz A, Szakos A, Hassan Z, Omazic B, Aschan J, Barkholt L, Le Blanc K. Mesenchymal stem cells for treatment of therapy-resistant graft-versus-host disease. Transplantation. 2006 May 27;81(10):1390-7. doi: 10.1097/01.tp.0000214462.63943.14. PMID 16732175